CLINICAL TRIAL: NCT04117087
Title: Pooled Mutant KRAS-Targeted Long Peptide Vaccine Combined With Nivolumab and Ipilimumab for Patients With Resected MMR-p Colorectal and Pancreatic Cancer
Brief Title: Pooled Mutant KRAS-Targeted Long Peptide Vaccine Combined With Nivolumab and Ipilimumab for Patients With Resected Mismatch Repair Protein (MMR-p) Colorectal and Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry); National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1994; IRB00210915 (Other: Johns Hopkins Medical Institution); 5P01CA247886 (NIH); K08CA248624 (NIH)
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer; Pancreatic Cancer
Keywords: KRAS Peptide Vaccine; Nivolumab; Ipilimumab; Anti-PD-1; Anti-CTLA-4; Neoantigen Vaccines; Cancer Vaccines; Immunotherapy; Colon Cancer; Pancreatic Ductal Adenocarcinoma (PDAC); Resected MMR-p Colorectal Cancer; Resected MMR-p Pancreatic Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms | interventions — poly ICLC; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Phase (Experimental): KRAS Vaccine Peptide, Nivolumab and Ipilimumab
  Interventions: Drug: KRAS peptide vaccine; Drug: Nivolumab; Drug: Ipilimumab
- Reinduction Treatment Phase (Experimental): KRAS Vaccine Peptide, Nivolumab and Ipilimumab
  Interventions: Drug: KRAS peptide vaccine; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: KRAS peptide vaccine — 1. KRAS peptide vaccine will be administered on cycle 1 (days 1, 8, 15) and R-Cycle 2 Day 1 (R-C2D1). Boost vaccinations with will be administered every 28 days at Reinduction cycle 5, 7, 9, 13. Extended vaccinations will be administered on Reinduction cycles 15 to 18, 19 and beyond (180 days ± 30 days for a total of 5 years on study.
  2. Drug: up to 1.8 mg KRAS peptide vaccine + 0.5mg Poly-ICLC
  Other Names: Hiltonol® (Poly-ICLC)
Drug: Nivolumab — 1. Nivolumab will be administered as a 30 minute IV infusion (-10min/+15min) on Day 1 of each 21 day cycle. Boost Phase will be administered every 28 days on cycles 5 thru 14.
  2. Drug: 3mg/kg IV, 480 mg IV
  Other Names: OPDIVO
Drug: Ipilimumab — 1. Ipilimumab (1 mg/kg) will be administered as a 30 minute IV infusion (-10min/+15min) on Day 1 of Cycles 1 and 3 of the study.
  2. Drug: 1mg/kg IV
  Other Names: YERVOY®

SUMMARY:
Phase 1 study for patients with resected PDAC after neoadjuvant and/ or adjuvant chemotherapy and/or radiation, as well as patients with metastatic colorectal cancer who have exposure to 2 or more lines of chemotherapy, to evaluate safety and the immune response to pooled mutant-KRAS peptide vaccine (KRAS peptide vaccine) with poly-ICLC adjuvant in combination with nivolumab and ipilimumab.

ELIGIBILITY:
Inclusion Criteria:

PDAC or metastatic MSS CRC Cohort:

* Have histologically or cytologically - proven cancer of the pancreas (PDA) or MSS colorectal (CRC) in one of the following categories:

  * PDAC must have no evidence of disease and last dose of neoadjuvant and/or adjuvant chemotherapy/radiation therapy/or surgery must be < 6 months from study entry.
  * Metastatic MSS CRC after exposure to 2 more lines of chemotherapy in the metastatic setting including 5-flurouracil, irinotecan, and oxaliplatin exposure. Patients treated with FOLFOXIRI may enroll after progression or intolerance to that regimen.
* For metastatic MSS CRC cohort, must have tumor lesions amenable to repeated biopsy, and patient's acceptance to have a tumor biopsy of an accessible lesion at baseline and on treatment if the lesion can be biopsied with acceptable clinical risk (as judged by the Principal Investigator).
* For metastatic MSS CRC patients, must have measurable disease per RECIST 1.1.

Reinduction Treatment Cohort:

* Have a single site of locoregional recurrence or distant metastasis noted on imaging > 12 months after the first dose of the mutant KRAS peptide vaccine with poly-ICLC adjuvant.
* Have completed definitive treatment for solitary recurrence per standard-of-care (e.g. surgical resection, radiation, and/or chemotherapy) <6 months prior to screening for reinduction treatment.

Both Cohorts:

*Age ≥18 years.

* Have sufficient archival tumor tissue for next-generation sequencing (NGS) and immune-phenotyping.
* Have one of the KRAS mutations included in the vaccine at the time of vaccination expressed in tumor.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Life expectancy of greater than 6 months.
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests prior to initial study drug.
* Woman of childbearing potential must have a negative pregnancy test and follow contraceptive guidelines as defined per protocol.
* Men must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria

* If expected to require any other form of systemic or localized antineoplastic therapy while on study.
* Within 2 weeks prior to first dose of study drug.

  * Systemic or topical steroids corticosteroids at immunosuppressive doses (> 10 mg/day of prednisone or equivalent). Inhaled or topical steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
  * Any palliative or adjuvant radiation or gamma knife radiosurgery.
  * Any chemotherapy.
* Within 4 weeks prior to first dose of study drug.

  * Any investigational cytotoxic drug.
  * Any investigational device.
  * Has received a live vaccine.
  * Received any allergen hyposensitization therapy.
  * Received any growth factors, e.g. granulocyte-colony stimulating factor (G-CSF), granulocyte macrophage-colony stimulating factor (GM-CSF), erythropoietin.
  * Any major surgery.
* PDAC or metastatic MSS CRC Cohort: Prior treatment with immunotherapy agents (including, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA4), etc.).
* Hypersensitivity reaction to any monoclonal antibody.
* Known history or evidence of brain metastases.
* Has active autoimmune disease that has required systemic treatment in the past 2 years, or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents.
* Known history or concurrent interstitial lung disease.
* Has a pulse oximetry < 92% on room air.
* Requires the use of home oxygen.
* Infection with HIV or hepatitis B or C.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, metastatic cancer, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has been diagnosed with another cancer or myeloproliferative disorder within the past 5 year.
* Has a diagnosis of immunodeficiency.
* Presence of any tissue or organ allograft, regardless of need for immunosuppression, including corneal allograft. Patients with a history of allogeneic hematopoietic stem cell transplant will be excluded.
* Any other sound medical, psychiatric, and/or social reason as determined by the Investigator.
* Unwilling or unable to follow the study schedule for any reason.
* Are pregnant or breastfeeding.
* For metastatic MSS CRC and Reinduction Treatment Cohorts, any peritoneal involvement by the tumor.
* For metastatic MSS CRC and Reinduction Treatment Cohorts, any radiological or clinical pleural effusions or ascites.
* For metastatic MSS CRC and Reinduction Treatment Cohorts, patients on parenteral nutrition.
* For metastatic MSS CRC and Reinduction Treatment Cohorts, patients with any single liver metastases greater than 5 cm or greater > 50% liver involvement.
* For metastatic MSS CRC and Reinduction Treatment Cohorts, history of malignant bowel obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing study drug-related toxicities | 2 years
  Number of participants experiencing study drug-related adverse events Grade 3 or higher as defined by CTCAE v5.0
Fold change in interferon-producing mutant-KRAS-specific cytotoxic (CD8) and helper (CD4) T cells at 16 weeks | Baseline, 16 weeks
  Evaluated by the fold change in interferon-producing mutant-KRAS-specific CD8 and CD4 T cells after vaccination at 16 weeks compare to pre-vaccination baseline.

SECONDARY OUTCOMES:
Disease Free Survival (DFS) | 4 years
  DFS is defined as the number of months from cycle 1, day 1 of vaccination until the first documented disease recurrence or death due to any cause in patients with resected PDAC. Will be censored at the date of the last progressive disease evaluation if no event observed.
Percentage change of interferon (IFN)-γ-producing mutant-KRAS-specific CD8 and CD4 T cells | 2 years
  Percent change of IFN-γ-producing mutant-KRAS-specific CD8 and CD4 T cells at any time after vaccination.
Objective Response Rate (ORR) per RECIST 1.1 | 4 years
  ORR is defined as the number of patients with metastatic microsatellite stable (MSS) CRC who are administered at least one dose of KRAS achieving a complete response (CR) partial response (PR) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) at any time during the study. CR = disappearance of all target lesions, PR is =>30 percent decrease in sum of diameters of target lesions, progressive disease (PD) is >20 percent increase in sum of diameters of target lesions, stable disease (SD) is <30 percent decrease or <20 percent increase in sum of diameters of target lesions.
Progression-free Survival (PFS) for RECIST 1.1 | 4 years
  PFS is defined as the numbers of months from the date of the first vaccine dose to the date of disease progression or death due to any cause, which ever occurs first, for Metastatic Colorectal Cancer (mCRC) patients. Censored at the date of last scan for subjects without documentation of disease progression (PD) at the time of analysis or relapse from complete response [CR] as assessed using RECIST 1.1 criteria) or death due to any cause. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30 percent decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20 percent increase in sum of diameters of target lesions, Stable Disease (SD) is <30 percent decrease or <20 percent increase in sum of diameters of target lesions.
Overall Survival (OS) | 4 years
  OS will be measured as the number of months from the date of first vaccine dose until death or end of follow up. OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis. Estimation based on the Kaplan Meier Curve

CONTACTS AND LOCATIONS:
Overall Officials: Nilofer Azad, MD, Principal Investigator — Johns Hopkins Medical Institution
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huff AL, Haldar SD, Gergis AA, Wang HH, Danilova L, Heumann T, Berg M, Wang Y, Andaloori L, Hernandez A, Longway G, Barrett B, Zhu Z, Davis-Marcisak E, Thoburn C, Leatherman J, Mitchell S, Lee JW, Shu DH, Konig MF, Mog BJ, Montagne J, Coyne EM, Bever K, Baretti M, Yarchoan M, Anders RA, Kagohara LT, Laheru D, Thomas AM, Durham J, Nauroth JM, Lu J, Wang H, Fertig EJ, Ho WJ, Azad NS, Jaffee EM, Zaidi N. Mutant KRAS vaccine with dual checkpoint blockade in resected pancreatic cancer: a phase I trial. Nat Commun. 2026 Feb 10;17(1):1538. doi: 10.1038/s41467-026-68324-4. PMID 41667470